CLINICAL TRIAL: NCT05068336
Title: Comparison of the Effects of Sevoflurane and Desflurane on Endothelial Glycocalyx in Laparoscopic Hysterectomy Surgery
Brief Title: Comparison of the Effects of Sevoflurane and Desflurane on Endothelial Glycocalyx
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, medical doctor, Kocaeli Derince Education and Research Hospital
Other Study IDs: 514-192-32
Record Dates: First submitted 2021-08-20; First posted 2021-10-05 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- desflurane: Anesthesia maintenance of the first group will be provided with desflurane, one of the inhalation anesthetics we routinely use. Before and after the operation, blood will be taken from the patients, and the blood will be centrifuged to evaluate the heparan sulfate and syndecan levels.
  Interventions: Diagnostic Test: desflurane anesthesia
- sevoflurane: Anesthesia maintenance of the first group will be provided with sevoflurane, one of the inhalation anesthetics we routinely use. Before and after the operation, blood will be taken from the patients, and the blood will be centrifuged to evaluate the heparan sulfate and syndecan levels.
  Interventions: Diagnostic Test: sevoflurane anesthesia

INTERVENTIONS:
Diagnostic Test: desflurane anesthesia — Anesthesia maintenance of the first group will be provided with desflurane, one of the inhalation anesthetics we routinely use. Before and after the operation, blood will be taken from the patients, and the blood will be centrifuged to evaluate the heparan sulfate and syndecan levels.
  Groups: desflurane
Diagnostic Test: sevoflurane anesthesia — Anesthesia maintenance of the first group will be provided with sevoflurane, one of the inhalation anesthetics we routinely use. Before and after the operation, blood will be taken from the patients, and the blood will be centrifuged to evaluate the heparan sulfate and syndecan levels.
  Groups: sevoflurane

SUMMARY:
The glycocalyx is a dynamic and complex biochemical structure composed of proteoglycans, glycoproteins, and soluble proteins. The glycocalyx interacts with various proteins such as albumin and orosomucoid to form a thick surface layer on the vessel surface that is physiologically active. This is called the endothelial surface layer. This structure is constantly changing with the blood flowing in the vein. The glycocalyx regulates oncotic pressure and also prevents leukocyte and platelet adhesion to the endothelium. Endothelial cell dysfunction is a valuable marker of increased vascular permeability and impaired angiogenesis due to cardiovascular, thoracic, renal, and metabolic diseases.

DETAILED DESCRIPTION:
The glycocalyx is a dynamic and complex biochemical structure composed of proteoglycans, glycoproteins, and soluble proteins. The glycocalyx interacts with various proteins such as albumin and orosomucoid to form a thick surface layer on the vessel surface that is physiologically active. This is called the endothelial surface layer. This structure is constantly changing with the blood flowing in the vein. The glycocalyx regulates oncotic pressure and also prevents leukocyte and platelet adhesion to the endothelium. Endothelial cell dysfunction is a valuable marker of increased vascular permeability and impaired angiogenesis due to cardiovascular, thoracic, renal, and metabolic diseases.

Some medical approaches, including anti-thrombin III, nitric oxide, the TNF-α analog etanercept, and inhalation agents, can repair or prevent deterioration of the endothelial glycocalyx. In a study by Chen et al., it was shown that Sevoflurane has a protective effect on syndecan and heparan sulfate, which are located in the glycocalyx structure, thus reducing leukocyte and platelet adhesion and protecting the vascular endothelium (8).

Kim et al. In a study conducted, it was shown that the protective effect of propofol, an intravenous anesthetic, on the vascular endothelium was greater than that of sevoflurane In our research, no study was found on the effect of another inhalation anesthetic, desflurane, on the vascular glycocalyx structure. In this study, we aimed to investigate and compare the effects of sevoflurane and desflurane on glycocalyx.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 18-65 age rang
* Being in the ASA 1-3 risk group
* patients receiving general anesthesia

Exclusion Criteria:

* refuse to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
glycocalyx components | the study will comlete in one month
  The primary aim of the study was to measure the levels of heparan sulfate and syndecan, which are markers of endothelial glycocalyx structure, after the use of desflurane or sevoflurane. High biomarker levels are associated with impaired glycocalyx structure

SECONDARY OUTCOMES:
haemodynamic changes | studdy will complete in one month
  The secondary aim of the study is to compare the hemodynamic effects of sevoflurane and desflurane.

CONTACTS AND LOCATIONS:
Locations (1):
- Tahsin Şimşek, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided